CLINICAL TRIAL: NCT03870607
Title: A Randomized Phase II Study of the Administration of Prebiotics and Probiotics During Definitive Treatment With Chemotherapy-radiotherapy for Patients With Squamous Cell Carcinoma of the Anal Canal (BISQUIT)
Brief Title: Prebiotics and Probiotics During Definitive Treatment With Chemotherapy-radiotherapy SCC of the Anal Canal (BISQUIT)
Acronym: BISQUIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Riechelmann, Head of Departament of Clinical Oncology, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2625-18
Record Dates: First submitted 2019-02-12; First posted 2019-03-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Anal Cancer Squamous Cell
Keywords: probiotics; prebiotics; microbiome
MeSH Terms: conditions — Anus Neoplasms | interventions — Prebiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Eligible patients who consent to participate in this study will be randomized 1: 1 in two groups: Group A or experimental and Group B or control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers will identify the patients through a unique number and through the initials of the name. Randomization will be simple and conducted independently by clinical trial support staff who are not participating in the study. The random sequence will be generated by computer program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotics and probiotics group (Experimental): This group will receive standard nutritional guidance from the institutional routine and prebiotics in combination with probiotics, starting one week before the start of Ch-RT and daily throughout the treatment up to 6 to 8 weeks post Ch-RT at the time of evaluation response (primary outcome).
  Interventions: Dietary Supplement: prebiotics in combination with probiotics
- Control group (No Intervention): This group will lead nutritionally based just before starting Ch-RT.

INTERVENTIONS:
Dietary Supplement: prebiotics in combination with probiotics — Administration of prebiotics in combination with probiotics before the start of Ch-RT
  Other Names: Symbioflor
  Arms: Prebiotics and probiotics group

SUMMARY:
Phase II randomized study of the use of pre-and probiotics during the definitive treatment of chemotherapy-radiotherapy (Ch-RT) for patients with localized anal canal squamous cell cancer (ACSCC) with the objective of increasing the effectiveness of conventional treatment based on the assumptions of that there is a need for research that increases the cure rates of the definitive treatment of Ch-RT in the ACSCC; ACSCC is a virus-associated tumor in many cases and therefore potentially immunogenic; immunotherapy is a promising strategy in ACSCC; and that pre- and probiotics can stimulate the immune system through modulation of the intestinal microbiota, and improve oncological outcomes.

DETAILED DESCRIPTION:
Although anal canal squamous cell carcinoma (ACSCC) is rare in developed countries, it has shown an annual increase of 4% in its incidence in Brazil, and according to data from the Oncocenter Foundation of São Paulo (FOSP), 2,338 cases were diagnosed in 2000 and 2016.

The standard treatment for localized ACSCC (without distant metastases) is definitive chemo-radiotherapy (Ch-RT) concomitant with administration of a fluoropyrimidine (5FU or capecitabine) combined with mitomycin or cisplatin, which provides cure rates of 60-80 % depending on the staging. When there is no complete remission, surgical rescue through anal amputation is the only potentially curative modality. However, this strategy is associated with great morbidity, besides negative emotional and social impacts, with consequent reduction of quality of life. Therefore, interventions that may increase the chance of cure in ACSCC should be investigated.

The main risk factors for ACSCC are human papillomavirus (HPV) infections and immunosuppression, including human immunodeficiency virus (HIV) infection. Chronic HPV infection and HIV-induced immunosuppression point to research strategies that strengthen the immune system to reduce the risk of developing ACSCC. In the metastatic setting, the use of immune checkpoint inhibitors, such as anti-programmed death protein-1 (PD1) antibodies, were shown to be promising in ACSCC patients, promoting response rates of approximately 25%. However, there is no evidence of modulation interventions of the immune system in patients with localized ACSCC.

Recently, studies have shown that the composition of the intestinal microbiota influences the onset of colorectal cancer, and may even disrupt the effects of chemotherapy in this neoplasm. A preclinical study in animal model showed that E. coli impaired the antitumor effect of fluoropyrimidines, drug used in colorectal cancer and ACSCC. The intestinal microbiota also participates in a large set of metabolic processes (such as reduction, hydrolysis, dehydroxylation, etc.) involved in drug metabolism. For example, some intestinal bacteria have β-glucuronidases that cleave glucuronide from the inactive metabolite of irinotecan (SN-38G), a drug used in gastrointestinal tumors, releasing active metabolite (SN38) in the intestine, causing diarrhea and colitis. Ciprofloxacin has been shown to inhibit this enzyme by suppressing the diarrhea associated with irinotecan in an experimental model of mice. Mycoplasma hyorhinis encodes a thymidine phosphorylase that strongly restricts the cytostatic activity of pyrimidine nucleoside analogues.

On the other hand, the replacement of the intestinal microbiota "carcinogenic" (Fusobacterium spp and Bacteriodes fragilis) by a protective microbiota (Bifidobacterium and Lactobacillus) has been the reason of numerous investigations with prebiotics and probiotics. According to the International Scientific Association of Probiotics and Prebiotics, probiotics are composed of living organisms which, when administered, promote health benefits, such as antimicrobial action against intestinal pathogens, modulation of the immune system, reduction of cholesterol levels, reduction of colitis and prevention of colorectal cancer. Kefir is an example of probiotic. Already prebiotics are inert ingredients that promote alteration in the composition or activity of the gastrointestinal microflora, conferring health benefits. Example of prebiotic is polysaccharide inulin. Studies with these compounds have been conducted, showing promising results. A small placebo-controlled trial using B. breve breve (Yakut®) in children undergoing chemotherapy for a variety of neoplasms has shown that this group had fewer episodes of fever and less frequency of use of intravenous antibiotics compared to controls. There are also studies that suggest that the alteration of the intestinal flora can increase the effectiveness of immunotherapy as a form of modulation of the immune system in several animal models of colorectal cancer. In addition, the use of this strategy could have a modulatory effect on local and systemic toxicity of the treatment, possibly reducing the morbidity of the treatment, as already suggested by studies in cervical carcinomas.

Despite the strong scientific rationale, there are no studies that have evaluated the use of probiotics or prebiotics in order to increase the effectiveness of conventional Ch-RT treatment in ACSCC. Therefore, based on the assumptions that there is a need for research that increases the cure rates of the definitive treatment of Ch-RT in ACSCC; ACSCC is a virus-associated tumor in many cases and therefore potentially immunogenic; immunotherapy is a promising strategy in ACSCC; and that pre- and probiotics can stimulate the immune system through modulation of the intestinal microbiota, and improve oncological outcomes, the investigators propose a randomized phase II study of the use of pre-probiotics during definitive treatment of Ch-RT for patients with ACSCC located.

The primary hypothesis of this study is that addition of pre- and probiotics increases the proportion of patients with complete clinical and radiological response after Ch-RT to ACSCC. Secondary hypotheses are that pre- and probiotics increase the metabolic response measured by positron emission computed tomography (PET-CT) with 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18-FDG) and promote greater control of local disease after Ch-RT; and reduce local and systemic toxicity of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years;
* Confirmed histological diagnosis of squamous cell carcinoma / squamous cell carcinoma of the anal canal (ACSCC);
* Patients with localized ACSCC (≥ T2N0M0, according to American Joint Committee on Cancer (AJCC) 8th edition) staged by conventional imaging methods according to institutional routine;
* Indication of starting definitive treatment with Ch-RT in the institution. HIV-positive patients may be included;
* Free and informed consent signed by the patient or legal representative

Exclusion Criteria:

* Diagnosis of perianal squamous cell carcinomas;
* Clinical condition leading to difficulty in swallowing;
* Patients with a contraindication to receiving Ch-RT, ie receiving only radiotherapy or not receiving polychemotherapy;
* Clinical condition that, due to the investigator's judgment, prevents adherence to the study
* Active infection requiring antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-03-13 (Actual); Primary Completion 2023-08-13 (Estimated); Study Completion 2024-02-11 (Estimated)

PRIMARY OUTCOMES:
Response rate (clinical and radiological) | Six to eight weeks from the end of Ch-RT
  absence of visible disease at the clinical examination and magnetic resonance imaging (MRI) of the pelvis (or pelvic tomography, if contraindicated to MRI) and without disease at a distance, through tomography of the chest and abdomen.

SECONDARY OUTCOMES:
Metabolic response by 18-FDG PET-CT | Six to eight weeks from the end of Ch-RT
  Comparing the mean pre-and post-Ch-RT volume-capture measurements of each patient at 6-8 weeks post Ch-RT
Complete clinical and radiological response rate | Six months
  defined as absence of disease visible to clinical and pelvic MRI (or pelvic tomography) exams and without disease at a distance, through tomography of the chest and abdomen;
Progression / disease free survival | through study completion, an average of 5 years
  defined as the time from day1 cycle 1 of Ch-RT treatment to local or remote relapse, or death from any cause, whichever occurs first.
Proportion of patients without colostomy | Twelve months
  Proportion of patients without colostomy 12 months after Ch-RT termination.
Incidence of Adverse Events Treatment-related | through study completion, an average of 5 years
  Adverse events of grade 2 or higher by the Common Adverse Event Toxicity Criteria (CTCAE) version 4.0.
Incidence of HPV in tumor tissue | through study completion, an average of 3 years
  Incidence of positivity for HPV screening in tumor tissue through genotyping
Variation of systemic immune parameters | through study completion, an average of 3 years
  Defined by variation in total number of lymphocytes, neutrophil / lymphocyte ratio (NLR) and lymphocyte / monocyte ratio (LMR)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel SP Riechelmann, MD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niederreiter L, Adolph TE, Tilg H. Food, microbiome and colorectal cancer. Dig Liver Dis. 2018 Jul;50(7):647-652. doi: 10.1016/j.dld.2018.03.030. Epub 2018 Apr 3. PMID 29705028
- [Background] Scott TA, Quintaneiro LM, Norvaisas P, Lui PP, Wilson MP, Leung KY, Herrera-Dominguez L, Sudiwala S, Pessia A, Clayton PT, Bryson K, Velagapudi V, Mills PB, Typas A, Greene NDE, Cabreiro F. Host-Microbe Co-metabolism Dictates Cancer Drug Efficacy in C. elegans. Cell. 2017 Apr 20;169(3):442-456.e18. doi: 10.1016/j.cell.2017.03.040. PMID 28431245
- [Background] Alexander JL, Wilson ID, Teare J, Marchesi JR, Nicholson JK, Kinross JM. Gut microbiota modulation of chemotherapy efficacy and toxicity. Nat Rev Gastroenterol Hepatol. 2017 Jun;14(6):356-365. doi: 10.1038/nrgastro.2017.20. Epub 2017 Mar 8. PMID 28270698
- [Background] Zou S, Fang L, Lee MH. Dysbiosis of gut microbiota in promoting the development of colorectal cancer. Gastroenterol Rep (Oxf). 2018 Feb;6(1):1-12. doi: 10.1093/gastro/gox031. Epub 2017 Oct 11. PMID 29479437
- [Background] Gopalakrishnan V, Helmink BA, Spencer CN, Reuben A, Wargo JA. The Influence of the Gut Microbiome on Cancer, Immunity, and Cancer Immunotherapy. Cancer Cell. 2018 Apr 9;33(4):570-580. doi: 10.1016/j.ccell.2018.03.015. PMID 29634945
- [Background] Ferreira MR, Muls A, Dearnaley DP, Andreyev HJ. Microbiota and radiation-induced bowel toxicity: lessons from inflammatory bowel disease for the radiation oncologist. Lancet Oncol. 2014 Mar;15(3):e139-47. doi: 10.1016/S1470-2045(13)70504-7. PMID 24599929
- [Result] de Souza DL, Curado MP, Bernal MM, Jerez-Roig J, Boffetta P. Mortality trends and prediction of HPV-related cancers in Brazil. Eur J Cancer Prev. 2013 Jul;22(4):380-7. doi: 10.1097/CEJ.0b013e32835b6a43. PMID 23238584
- [Result] Morris VK, Salem ME, Nimeiri H, Iqbal S, Singh P, Ciombor K, Polite B, Deming D, Chan E, Wade JL, Xiao L, Bekaii-Saab T, Vence L, Blando J, Mahvash A, Foo WC, Ohaji C, Pasia M, Bland G, Ohinata A, Rogers J, Mehdizadeh A, Banks K, Lanman R, Wolff RA, Streicher H, Allison J, Sharma P, Eng C. Nivolumab for previously treated unresectable metastatic anal cancer (NCI9673): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Apr;18(4):446-453. doi: 10.1016/S1470-2045(17)30104-3. Epub 2017 Feb 18. PMID 28223062
- [Result] James RD, Glynne-Jones R, Meadows HM, Cunningham D, Myint AS, Saunders MP, Maughan T, McDonald A, Essapen S, Leslie M, Falk S, Wilson C, Gollins S, Begum R, Ledermann J, Kadalayil L, Sebag-Montefiore D. Mitomycin or cisplatin chemoradiation with or without maintenance chemotherapy for treatment of squamous-cell carcinoma of the anus (ACT II): a randomised, phase 3, open-label, 2 x 2 factorial trial. Lancet Oncol. 2013 May;14(6):516-24. doi: 10.1016/S1470-2045(13)70086-X. Epub 2013 Apr 9. PMID 23578724
- [Result] Ambalam P, Raman M, Purama RK, Doble M. Probiotics, prebiotics and colorectal cancer prevention. Best Pract Res Clin Gastroenterol. 2016 Feb;30(1):119-31. doi: 10.1016/j.bpg.2016.02.009. Epub 2016 Feb 19. PMID 27048903
- [Result] Braghiroli MI, Mota JM, Duarte PS, Morita TO, Bariani GM, Nebuloni D, Buchpiguel CA, Hoff PM, Riechelmann RP. Evaluation of 18F-FDG PET-CT as a prognostic marker in advanced biliary tract cancer. Nucl Med Commun. 2018 Mar;39(3):252-259. doi: 10.1097/MNM.0000000000000810. PMID 29381586

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03870607/Prot_SAP_ICF_000.pdf